CLINICAL TRIAL: NCT07243561
Title: Prospective Clinical Study on Human Umbilical Cord Mesenchymal Stem Cell-Derived Exosomes for the Treatment of Childhood Autism
Acronym: EXO-ASD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dongfang People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-DFKYLL-002
Record Dates: First submitted 2025-11-13; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder (ASD; Prospective Study
Keywords: Autism Spectrum Disorder; umbilical cord mesenchymal stem cells; exosome
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hUC-MSC-EXOs Nasal Spray Group (Experimental)
  Interventions: Biological: hUC-MSC-Exos Nasal Spray
- No-Intervention Control Group (No Intervention)

INTERVENTIONS:
Biological: hUC-MSC-Exos Nasal Spray — The total therapeutic dosage is set at 400 billion hUC-MSC-EXOs particles. Each nasal administration delivers 40 billion particles, with a total of 10 administrations completing the full course. The treatment is administered on an alternate-day schedule.
  Arms: hUC-MSC-EXOs Nasal Spray Group

SUMMARY:
This clinical study aims to evaluate whether a nasal spray containing exosomes derived from human umbilical cord mesenchymal stem cells (hUC-MSC-EXOs) can safely and effectively improve core symptoms in children aged 3-7 years with autism spectrum disorder (ASD). It is a 24-week, randomized, controlled, open-label trial. Forty pediatric patients with ASD will be randomly assigned at a 1:1 ratio to two groups: an active exosome nasal spray treatment group and a no-intervention control group. The treatment group will receive the nasal spray every other day, totaling 10 administrations throughout the study. The no-intervention control group will receive no experimental treatment but will undergo the same assessments and safety checks concurrently with the treatment group. This design aims to monitor the safety and efficacy of the hUC-MSC-EXOs nasal spray.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis meets the ICD-11 ASD criteria or DSM-5 ASD clinical diagnostic standards.
* No significant improvement in core symptoms was observed after ≥3 months of standardized behavioral intervention.
* Score ≥30 on the CARS2, indicating mild-to-moderate or more severe autism.
* Aged 3 (inclusive) to 7 (inclusive) years, regardless of gender
* Voluntary participation in this clinical study, with written informed consent provided by the patient's legal guardian, and willingness to undergo examinations, treatment, and cooperate with follow-up visits.
* In the investigator's judgment, the patient is capable of understanding and complying with study requirements.

Exclusion Criteria:

* History of severe allergic reactions.
* Any severe mental disorder or other types of autism spectrum disorders.
* History of epileptic seizures within the past six months.
* Autism secondary to epilepsy, cerebrovascular disease, or traumatic brain injury.
* Disease severity rated as normal, borderline mental disorder, or mild mental disorder on the Clinical Global Impression scale.
* Moderate or severe extrapyramidal symptoms or tardive dyskinesia.
* Severe self-injurious behavior.
* Active systemic or severe localized infections, including human immunodeficiency virus, syphilis, and hepatitis.
* Autoimmune diseases.
* Major organ impairment.
* Severe pulmonary or hematological diseases, malignancies, or immunodeficiency.
* Concurrent treatments that may interfere with the safety and efficacy evaluation of stem cell therapy.
* Participation in other clinical trials within the past three months.
* Other clinical conditions deemed by investigators as unsuitable for study inclusion.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events | Week 2, Week 6, Week 24
  The incidence of treatment-related adverse events will be assessed and graded according to the Common Terminology Criteria for Adverse Events version 5.0. The number of participants experiencing any treatment-related adverse event will be recorded and reported.
Childhood Autism Rating Scale, Second Edition (CARS-2) Score | Week 6, Week 24
  Scale Description: The CARS-2 is a 15-item behavior rating scale used to diagnose and assess the severity of ASD.
  Range of Scores: 15 to 60. Interpretation: A higher score indicates a worse outcome.

SECONDARY OUTCOMES:
Autism Behavior Checklist (ABC) | Week 6, Week 24
  Scale Description: The ABC is a 57-item checklist used to screen for and assess behaviors associated with ASD.
  Range of Scores: 0 to 158. Interpretation: A higher score indicates a worse outcome.
Serum Level of Tumor Necrosis Factor-Alpha (TNF-α) | Week 6, Week 24
  Serum concentration of the inflammatory cytokine TNF-α. The unit of measure is pg/mL.

CONTACTS AND LOCATIONS:
Locations (1):
- Dongfang People's Hospital, Dongfang, Hainan, China

IPD SHARING:
Plan to Share IPD: No